CLINICAL TRIAL: NCT05681884
Title: Faricimab for Retinal Non-Perfusion Associated With Non-Proliferative Diabetic Retinopathy: The MAGIC Phase 2, Multi-Center, Open-Label, Randomized Controlled Trial
Brief Title: Safety and Efficacy of Faricimab in Patients With NPDR
Acronym: MAGIC
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Greater Houston Retina Research (Other)
Collaborators: Genentech, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ML43601; 164104 (Other: FDA (IND))
Record Dates: First submitted 2022-11-04; First posted 2023-01-12 (Actual); Last update posted 2025-01-24 (Actual); Status verified 2025-01

CONDITIONS: Non-Proliferative Diabetic Retinopathy
MeSH Terms: interventions — faricimab

STUDY DESIGN:
Intervention Model Description: Randomized during the enrollment phase of the study in a 1:1 ratio to one of two treatment arms.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Group 1 (Experimental): Subjects will be administered intravitreal faricimab 6 mg every 4 weeks (defined as every 28 days + 7 days and at least 21 days between injections) through week 48. Starting at Week 48, subjects will be treated every 16 weeks (weeks 48, 64 & 80) with an end of study visit at week 96.
  Rescue: At any visit after Week 48, if rescue criteria are met, faricimab 6mg will be given every 4 weeks and the subject will continue dosing through the end of the trial.
  Interventions: Drug: Faricimab
- Group 2 (Experimental): Subjects are seen and observed every 16 weeks. Starting at Week 48, subjects will be administered intravitreal faricimab 6 mg every 4 weeks from week 48 to week 92, (defined as every 28 days ± 7 days and at least 21 days between injections) with an end of study visit at week 96.
  Rescue: At any visit before Week 48, if rescue criteria are met, faricimab 6mg will be given every 4 weeks and the subject will continue dosing through the end of the trial.
  Interventions: Drug: Faricimab

INTERVENTIONS:
Drug: Faricimab — Faricimab is a humanized bispecific antibody binding to human Ang-2 and VEGF. For Phase III studies, the Ro 686-7461 drug product is provided in single-dose 2-mL glass vials (6 mg/0.05 mL) with L-histidine/acetate buffered solution (approximately pH 5.5) containing sodium chloride, sucrose, L-methionine, polysorbate 20, and water for injection.

SUMMARY:
The purpose of this Phase 2 study is comprised of two groups to evaluate the safety, tolerability, and efficacy of faricimab in patients with Non-Proliferative Diabetic Retinopathy.

DETAILED DESCRIPTION:
Group 1: Subjects will be administered intravitreal faricimab every 4 through week 48 and then will be receive faricimab every 16 weeks with an end of study visit at week 96. At any visit after Week 48, if rescue criteria are met, faricimab 6mg will be given every 4 weeks and the subject will continue dosing through the end of the trial.

Group 2: Subjects are seen and observed every 16 weeks. Starting at Week 48, subjects will be administered intravitreal faricimab every 4 weeks from week 48 to week 92 with an end of study visit at week 96. At any visit before Week 48, if rescue criteria are met, faricimab will be given every 4 weeks and the subject will continue dosing through the end of the trial.

ELIGIBILITY:
Inclusion Criteria:

* Provide signed IRB-approved informed consent form (ICF) prior to any study-specific procedures
* Willing and able to comply with clinic visits and study-related procedures and likely to return for all study visits, in the investigator's judgement
* Men or women > 18 years of age at the time of signing the Informed Consent Form
* Diagnosis of diabetes mellitus (type 1 or type 2)
* For women of childbearing potential: agreement to remain abstinent (refrain from heterosexual intercourse) or use acceptable contraceptive methods that result in a failure rate of < 1% per year during the treatment period and for at least 3 months after the final dose of study treatment. A woman is considered to be of childbearing potential if she is post-menarcheal, has not reached a post-menopausal state (>12 continuous months of amenorrhea with no identified cause other than menopause), and has not undergone surgical sterilization (removal of ovaries and/or uterus). The definition of childbearing potential may be adapted for alignment with local guidelines or requirements. Examples of acceptable contraceptive methods include bilateral tubal ligation, male sterilization, hormonal contraceptives that inhibit ovulation, hormone-releasing intrauterine devices, and copper intrauterine devices.

Contraception methods that do not result in a failure rate of < 1% per year such as male or female condom with or without spermicide; and cap, diaphragm, or sponge with spermicide are not acceptable.

The reliability of sexual abstinence should be evaluated in relation to the duration of the clinical trial and the preferred and usual lifestyle of the subject. If a subject is usually not sexually active but becomes active, they, with their partner, must comply with the contraceptive requirements of the study.

Ocular inclusion criteria for study eye:

Subjects must meet the following ocular inclusion criteria for the study eye for entry into the study:

* ETDRS BCVA > 20/400 in the study eye
* Non-proliferative diabetic retinopathy, as confirmed by the site investigator
* Substantial non-perfusion (defined as greater than 5 disc areas on Wide-Field Fluorescein Angiograph (WFFA)), as assessed by site investigator

Exclusion Criteria:

* Any known hypersensitivity to any of the components in the faricimab injection
* Any known hypersensitivity to any contrast media (e.g., fluorescein), dilating eye drops, disinfectants (e.g., iodine), or any of the anesthetics and antimicrobial preparations used by the site during the study
* Active cancer within the past 12 months prior to Screen/Baseline except for appropriately treated carcinoma in situ of the cervix, non-melanoma skin carcinoma, and prostate cancer with a Gleason score of ≤6 and a stable prostate-specific antigen for >12 months
* Stroke (cerebral vascular accident) or myocardial infarction within 6 months prior to Screen/Baseline
* Pregnant or breastfeeding, or intending to become pregnant during the study or within 3 months after the final dose of faricimab

  o Women of childbearing potential must have a negative urine pregnancy test at the Screen/Baseline visit for both Group 1 and Group 2. Women of childbearing potential must also have a negative urine pregnancy test on any visit where they will receive treatment with IP or rescue medication. Urine pregnancy tests must be completed prior to the administration of IP/rescue medication and prior to FA being performed.
* Participation in an investigational trial that involves treatment with any drug or device (with the exception of vitamins or minerals) within 3 months (or 5 half-lives, whichever is longer) prior to Screen/Baseline, or during the course of this study
* Any prior or concomitant systemic anti-VEGF treatment within 4 months prior to Screen/Baseline
* Any use of any prohibited therapies during times of prohibition.

Ocular exclusion criteria for study eye:

Subjects who meet any of the following exclusion criteria for the study eye will be excluded from study entry:

* Any history of treatment with anti-VEGF or any periocular or IVT corticosteroids in the study eye within 4 months prior to Screen/Baseline
* SD-OCT central subfield thickness (CST) measurement > 325 µm, in the study eye due to DME.
* Evidence of infectious ocular infection, in the study eye at Screen/Baseline
* Any pan-retinal photocoagulation (PRP) treatment received in the study eye prior to Screen/Baseline
* Retinal vein occlusion in the study eye
* Cystoid macular edema not attributed to diabetes (instead caused by epiretinal membrane, macular telangiectasia, Coats disease, and inherited retinal diseases) in the study eye
* Current vitreous hemorrhage obscuring imaging in the study and/or dilated indirect examination
* Any intraocular surgery (e.g., cataract surgery) within 4 weeks prior to Screen/Baseline in the study eye
* Active intraocular inflammation including scleritis at screening/baseline

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 179 (Actual)
Dates: Start 2023-05-16 (Actual); Primary Completion 2026-03-20 (Estimated); Study Completion 2026-04-13 (Estimated)

PRIMARY OUTCOMES:
Primary Objective | 48 weeks
  Analyze the change in the area of retinal non-perfusion (RNP) within the macula over 48 weeks using ultrawide-field fluorescein angiography (UWFA) within eyes that have NPDR.
Primary Objective | 48 weeks
  Analyze the change in the area of retinal non-perfusion (RNP) outside the macula over 48 weeks using ultrawide-field fluorescein angiography (UWFA) within eyes that have NPDR.

SECONDARY OUTCOMES:
Change in area of RNP | Baseline through week 96
  Change in area of RNP, as assessed by a central reading center; linear regression of change in area of RNP (dependent variable) between the monthly faricimab and observation groups, adjusted for age, sex, and disease severity as defined by Baseline ETDRS
Change in area of RNP within the macula | Baseline through week 48 and from baseline through week 96
  Change in area of RNP within the macula, as assessed by ultrawide-field fluorescein; linear regression of change in area of RNP (dependent variable) between the monthly faricimab and observation groups, adjusted for age, sex, and disease severity as defined by Baseline ETDRS
Change in area of RNP outside of the macula | Baseline through week 48 and from baseline through week 96
  Change in area of RNP outside of the macula, as assessed by ultrawide-field fluorescein from baseline to week 96; linear regression of change in area of RNP (dependent variable) between the monthly faricimab and observation groups, adjusted for age, sex, and disease severity as defined by Baseline ETDRS
Percentage of subjects with disease | Baseline through week 96
  Percentage of subjects with neovascularization and/or vitreous hemorrhage and/or DME
Mean change in ETDRS | Baseline through week 48 and from baseline through week 96
  Mean change in ETDRS BCVA
Mean change in CST | Baseline through week 48 and from baseline through week 96
  Mean change in CST
Contrast Sensitivity | Baseline through Week 48 and from baseline through week 96
  Contrast sensitivity as measured using the quantitative Contrast Sensitivity Function (qCSF) testing on the Manifold Contrast Vision
Natural History of RNP | Baseline through Week 48 and from baseline through week 96
  Natural history of RNP through detection of apoptosing retinal cells (DoARC) imaging
2-step Improvement in DRSS | 48 weeks and 96 weeks
  Proportion of subjects with at least a 2-step improvement in DRSS

CONTACTS AND LOCATIONS:
Locations (16):
- United States (16):
  - California Retina Consultants, Bakersfield, California
  - Retinal Consultants Medical Group, Modesto, California
  - Florida Retina Institute, Orlando, Florida
  - Retina Group of Florida, Sarasota, Florida
  - Retina Consultants of Minnesota St. Louis Park, Saint Louis Park, Minnesota
  - Mississippi Retina Associates, Jackson, Mississippi
  - Long Island Vitreoretinal Consultants, Westbury, New York
  - North Carolina Retina Associates, Wake Forest, North Carolina
  - Charleston Neuroscience Institute, Ladson, South Carolina
  - Palmetto Retina Center, West Columbia, South Carolina
  - Austin Retina Associates, Austin, Texas
  - Retina Consultants of Texas, Beaumont, Texas
  - Retina Consultants of Texas, Bellaire, Texas
  - Retina Consultants of Texas, Katy, Texas
  - Retina Consultants of Texas, San Antonio, Texas
  - Retina Consultants of Texas, The Woodlands, Texas

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Zhou AW, Sahraravand RA, Baumann LM, Teagle GM, Brown J, Pieramici D, Holy SE, Borne MJ, Wong RW, Cunningham MA, Pearce WA, Rahman EZ, Chang M, Bhavsar AR, Brown DM, Alfaro DV, Fan KC, Cehofski LJ, Ip M, Sadda SR, Lesmes LA, Ehlers JP, Chaudhary V, Al-Khersan H, Wykoff CC. MAGIC: Study Design and Rationale for the Phase 2 Clinical Trial of Faricimab for Non-Proliferative Diabetic Retinopathy. Ophthalmologica. 2026 Jan 26:1-16. doi: 10.1159/000550491. Online ahead of print. PMID 41587134